CLINICAL TRIAL: NCT06540872
Title: Multimodal Imaging With FAPI-PET/MRI in Breast Carcinoma-In-Situ for Detection of Occult Invasive Cancer
Acronym: MI-CISDIR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universität Münster (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WWU22_0012; 2023-509860-47-00 (Other: EMA Clinical Trial Information System (EU CT number))
Record Dates: First submitted 2024-06-11; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma, Intraductal, Noninfiltrating
Keywords: breast cancer; PET/MRI; DCIS; ductal carcinoma in situ; FAPI
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — FAPI-46

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All participants receive the drug [68Ga]Ga-FAPI-46 and imaging
  Interventions: Drug: [68Ga]Ga-FAPI-46

INTERVENTIONS:
Drug: [68Ga]Ga-FAPI-46 — Participants receive the weakly radioactive drug [68Ga]Ga-FAPI-46 through their vein and lie in an imaging device (PET/MRI) for 30 minutes. After a break of 30 minutes, they will lie in the imaging device for another 15 minutes.
  Other Names: [68Ga]FAPI-46

SUMMARY:
DCIS (ductal carcinoma in situ) is a common pre-stage for breast cancer. The goal of this clinical trial is to learn if FAPI-PET/MRI (an imaging technique with a weakly radioactive drug) helps to diagnose hidden invasive breast cancer in participants with DCIS. The main question it aims to answer is:

How good can FAPI-PET/MRI diagnose hidden invasive breast cancer in DCIS?

Researchers will compare FAPI-PET/MRI results to tissue samples obtained from surgery treatment to see if the FAPI-PET/MRI images show invasive breast cancer certainly.

Participants will

* receive the radioactive drug and lie in an imaging device for 45 minutes including a break
* visit the clinic once again for a checkup and test

DETAILED DESCRIPTION:
Ductal carcinoma in situ (DCIS) is a common precursor to breast cancer where abnormal cells are present within the milk ducts without breaking through their walls (in situ). If these cancerous cells have already breached the boundaries of the milk ducts, it is referred to as "invasive carcinoma." About half of these precancerous conditions develop further into invasive carcinomas over time. However, since doctors cannot precisely predict this at an individual level, treating DCIS often involves removing the affected tissue to prevent progression towards invasive cancer. Typically, diagnosis relies on performing a biopsy, during which cells from the altered tissue are extracted and examined under a microscope. Unfortunately, determining whether or not an invasive carcinoma has developed is not always possible with certainty with this method; indeed, about one quarter of cases involving existing invasive carcinomas might remain undetected by conventional biopsy procedures.

Consequently, being able to ascertain before surgery if an invasive carcinoma exists or not would be highly beneficial. This study examines a novel method that could potentially enhance the discovery of hidden (also called 'occult') invasive carcinomas. Specifically, it employs positron emission tomography (PET) utilizing a radiopharmaceutical agent known as [68Ga]Ga-FAPI-46. This compound selectively targets and binds to fibroblast activation protein (FAP), abundant on surfaces of tumor-associated fibroblasts. By tagging this structure with a radiotracer, researchers aim to achieve precise visualization and assessment of tumor extent. For the PET examination, a minimal dose of the radiopharmaceutical is administered intravenously while sensitive cameras capture images of particular body sections externally (PET). Additionally, magnetic resonance imaging (MRI) of the breast is conducted concurrently to ensure anatomical orientation, image enhancement (attenuation correction), and additional information acquisition.

The trial visits will be scheduled during the regular treatment process. These will not extend the participant's overall treatment duration significantly, as all measures within the scope of the study typically occur within 30 days, but no more than 51 days. During this period, effective contraception is necessary.

Researchers will then compare the imaging results to the pathology ground truth to evaluate the feasibility of the method.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed DCIS with extent in mammography, MRI or ultrasound suspected to range > 4 cm
* Planned DCIS resection (breast conserving or mastectomy) as per guideline recommendation
* Written informed consent
* For women of child bearing potential: confirmed menstrual period (if applicable) and a negative highly sensitive urine or serum pregnancy test
* Women of childbearing potential (WOCBP) and male patients with partners of childbearing/reproductive potential must agree to use highly effective contraception (Pearl index < 1) when sexually active. This applies for the time period between signing of the informed consent form up to the final trial visit.

Exclusion Criteria:

* Contraindications for MRI (specific metallic implants, severe claustrophobia, history of anaphylaxis following MRI contrast agent application)
* GFR < 30 mL/(min∙1.73 m²)
* Current pregnancy or within last 8 weeks before begin of study participation
* Current nursing or within last 8 weeks before begin of study participation
* Inability to understand the nature, risks, and benefits of the study
* History of diagnosis of ipsilateral invasive breast cancer
* Concurrent diagnosis of contralateral invasive cancer, if not curatively treated by surgery > 1 year ago
* Known hypersensitivity to the active substance or to any of the excipients of the Investigational Medicinal Product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of feasibility of detection of occult invasive cancer in diagnosed DCIS of [68Ga]Ga-FAPI-46 breast PET/MRI | Within one year after end of trial
  Sensitivity based on blinded readers' PET/MRI visual assessment: "Suspicious for occult carcinoma: Yes/No"
Evaluation of feasibility of detection of occult invasive cancer in diagnosed DCIS of [68Ga]Ga-FAPI-46 breast PET/MRI | Within one year after end of trial
  Specificity based on blinded readers' PET/MRI visual assessment: "Suspicious for occult carcinoma: Yes/No"

SECONDARY OUTCOMES:
Evaluation of feasibility of detection of occult invasive cancer in diagnosed DCIS of [68Ga]Ga-FAPI-46 breast PET/MRI | Within one year after end of trial
  Optimal threshold based on tumor-to-background ratio of SUVmax (60-75min)
Evaluation of feasibility of detection of occult invasive cancer in diagnosed DCIS of [68Ga]Ga-FAPI-46 breast PET/MRI | Within one year after end of trial
  Area-under-the-curve of receiver-operating-characteristics curve based on tumor-to-background ratio of SUVmax (60-75min)
Diagnostic Odds Ratio (DOR) to evaluate possible superiority of PET/MRI visual assessment over breast MRI alone | Within one year after end of trial
  Based on Blinded readers' PET/MRI vs MRI only visual assessment: "Suspicious for occult carcinoma: Yes/No"
Evaluate the added value for diagnostic performance of MRI measures of diffusibility | Within one year after end of trial
  Sensitivity and specificity of lesion MRI diffusion weighted MRI apparent diffusion coefficient (ADC)
Evaluate the added value for diagnostic performance of MRI measures of perfusion and permeability | Within one year after end of trial
  Sensitivity and specificity of the DCE-MRI dynamic feature "Maximal Slope"
Evaluate the added value for diagnostic performance of MRI measures of perfusion and permeability | Within one year after end of trial
  Sensitivity and specificity of the DCE-MRI dynamic feature "Bolus arrival time"
Evaluate the added value for diagnostic performance of MRI measures of perfusion and permeability | Within one year after end of trial
  Sensitivity and specificity of the DCE-MRI pharmacokinetic modeling parameter: Volume transfer constant (KTrans)
Evaluate the added value for diagnostic performance of MRI measures of perfusion and permeability | Within one year after end of trial
  Sensitivity and specificity of the DCE-MRI pharmacokinetic modeling parameter: Fractional plasma volume (Vp)
Evaluate the diagnostic performance of the PET parameter SUVmax (60-75min) | Within one year after end of trial
  Sensitivity and specificity of static PET SUVmax (60-75min)
Evaluate the diagnostic performance of PET pharmacokinetic modeling parameters | Within one year after end of trial
  Sensitivity and specificity of dynamic PET pharmacokinetic modeling parameter binding potential (BP)
Evaluate impact of PET/MRI on follow-up minimal invasive diagnostic procedures | Within one year after end of trial
  Number of additional biopsies triggered by PET/MRI visual assessment
Evaluate impact of MRI on follow-up minimal invasive diagnostic procedures | Within one year after end of trial
  Number of additional biopsies triggered by MRI visual assessment
Evaluate the correspondence of FAP-expression determined by immunohistochemistry and PET | Joint analysis of the collected samples after the end of the trial. Samples were collected during regular surgery after the final trial visit.
  Correlation of immunohistopathology FAP visual staining score with SUVmax (60-75min)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Day of trial medication application and final visit (5-21 days after drug receival)
  Adverse events following [68Ga]Ga-FAPI-46 application

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Backhaus, Dr. med., Principal Investigator — Department of Nuclear Medicine, University Hospital Münster
Locations (2):
- Germany (2):
  - Department of Nuclear Medicine, University Hospital Essen, Essen, North Rhine-Westphalia
  - Department of Nuclear Medicine, University Hospital Münster, Münster, North Rhine-Westphalia